CLINICAL TRIAL: NCT05748691
Title: Trial of Switching High-sensitivity Cardiac Troponin Assays in Suspected Acute Coronary Syndrome: an Interrupted Time Series Analysis (TWITCH-ED Study)
Brief Title: Switching From Cardiac Troponin I to T
Acronym: TWITCH-ED
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: DL-2022-046
Record Dates: First submitted 2023-01-09; First posted 2023-03-01 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction; Acute Myocardial Ischemia; Myocardial Injury; Chest Pain; Heart Failure
Keywords: Acute Coronary Syndrome; Acute Myocardial Infarction; Myocardial Injury; High-Sensitivity Cardiac Troponin T; High-Sensitivity Cardiac Troponin I; Biomarker; Acute Cardiovascular Care; Diagnostic Pathways; Outcomes; Sex; Sex-specific Thresholds; Upper Reference Limits
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Heart Failure; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation group: Clinical use of hs-cTnI in patients with suspected acute coronary syndrome
- Post-implementation group: Clinical use of hs-cTnT in patients with suspected acute coronary syndrome
  Interventions: Diagnostic Test: Clinical implementation of hs-cTnT

INTERVENTIONS:
Diagnostic Test: Clinical implementation of hs-cTnT — To investigate the clinical impact on the transition from a hs-cTnI assay to a hs-cTnT assay in consecutive patients presenting to the Emergency Department or Acute Medical Unit with suspected acute coronary syndrome.
  Groups: Post-implementation group

SUMMARY:
Cardiac troponin is central to the diagnosis of myocardial infarction and high-sensitivity cardiac troponin (hs-cTn) assays are the preferred choice for the assessment of patients with suspected acute coronary syndrome.

Since the introduction of hs-cTn assays in Europe in 2010, most hospitals have switched from contemporary sensitive cardiac troponin assays to a hs-cTn assay. The implementation of hs-cTn assays has led to an increase in the number of patients identified with myocardial injury. Although both hs-cTnI and hs-cTnT assays are recommended in current guidelines, the impact of switching from a hs-cTnI assay to a hs-cTnT assay on clinical practice is unknown. At this point, no studies have evaluated the impact of implementing sex-specific hs-cTnT thresholds on the diagnosis of myocardial infarction and outcome in clinical practice.

The investigators propose to determine the proportion of patients with and without myocardial injury admitted to the hospital before and after implementation of a hs-cTnT assay and to evaluate the impact on investigations, care and clinical outcomes in consecutive patients with suspected acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Symptoms of possible acute coronary syndrome
* High-sensitivity cardiac troponin measured at presentation

Exclusion Criteria:

* Insufficient clinical information to perform record linkage
* Previous enrolment in the study
* Patients with ST-segment elevation myocardial infarction (STEMI)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to an Emergency Department or an Acute Medical Unit in NHS Lothian between October 25th 2020 and October 25th 2022 where the attending clinician measures cardiac troponin for suspected acute coronary syndrome will be identified by NHS Lothian staff or the research team using an existing screening tool embedded into the ordering of cardiac troponin testing.
  We will compare the clinical impact of two guideline recommended high-sensitivity cardiac troponin assays in routine health care. We will not seek individual patient consent as this is an evaluation of a change in routine clinical care using approved tests, there are no specific research procedures, and we wish to evaluate performance in those patients in whom clinicians apply the test to avoid selection bias.
Sampling Method: Probability Sample
Enrollment: 26000 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with suspected acute coronary syndrome admitted to hospital | Up to 24 hours
  To determine the proportion of patients with and without myocardial injury admitted to the hospital before and after implementation of the hs-cTnT assay

SECONDARY OUTCOMES:
Proportion of patients with myocardial injury admitted to hospital | Up to 24 hours
  To determine the proportion of patients with myocardial injury admitted to hospital
Length of hospital stay | Up to 30 days
  To determine the length of hospital stay
Clinical diagnosis of myocardial infarction | Up to 24 hours
  To determine the prevalence of myocardial infarction
Clinical diagnosis of heart failure | Up to 24 hours
  To determine the prevalence of heart failure
Coronary angiography during hospital admission | Up to 30 days
  To determine the number of coronary angiograms performed during hospital admission
Echocardiography during hospital admission | Up to 30 days
  To determine the number of echocardiograms performed during hospital admission
New prescription of evidence-based treatment for coronary artery disease or heart failure following discharge | Up to 30 days
  To determine the number of new prescriptions of evidence-based treatment for coronary artery disease or heart failure following discharge
Revascularization at 30 days and one year | 30 days and 1 year
  To determine the rate of coronary revascularization at 30 days and one year
Reattendance with suspected acute coronary syndrome at 30 days and one year | 30 days and 1 year
  To determine the rate of reattendance with suspected acute coronary syndrome at 30 days and one year
Subsequent myocardial infarction at 30 days and one year | 30 days and 1 year
  To determine the prevalence of subsequent myocardial infarction at 30 days and one year
Subsequent heart failure at 30 days and one year | 30 days and 1 year
  To determine the prevalence of subsequent heart failure at 30 days and one year
Subsequent myocardial infarction, heart failure or cardiovascular death at 30 days and one year | 30 days and 1 year
  To determine the prevalence of subsequent myocardial infarction, heart failure or cardiovascular death at 30 days and one year
Cardiovascular death at 30 days and one year | 30 days and 1 year
  To determine the prevalence of cardiovascular death at 30 days and one year
All-cause death at 30 days and one year | 30 days and 1 year
  To determine the prevalence of all-cause death at 30 days and one year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Shah ASV, Anand A, Strachan FE, Ferry AV, Lee KK, Chapman AR, Sandeman D, Stables CL, Adamson PD, Andrews JPM, Anwar MS, Hung J, Moss AJ, O'Brien R, Berry C, Findlay I, Walker S, Cruickshank A, Reid A, Gray A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Harkess R, Parker RA, Keerie C, Weir CJ, Mills NL; High-STEACS Investigators. High-sensitivity troponin in the evaluation of patients with suspected acute coronary syndrome: a stepped-wedge, cluster-randomised controlled trial. Lancet. 2018 Sep 15;392(10151):919-928. doi: 10.1016/S0140-6736(18)31923-8. Epub 2018 Aug 28. PMID 30170853
- [Background] Lee KK, Ferry AV, Anand A, Strachan FE, Chapman AR, Kimenai DM, Meex SJR, Berry C, Findlay I, Reid A, Cruickshank A, Gray A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Keerie C, Weir CJ, Shah ASV, Mills NL; High-STEACS Investigators. Sex-Specific Thresholds of High-Sensitivity Troponin in Patients With Suspected Acute Coronary Syndrome. J Am Coll Cardiol. 2019 Oct 22;74(16):2032-2043. doi: 10.1016/j.jacc.2019.07.082. PMID 31623760
- [Background] Mjoen G, Maggiore U, Kessaris N, Kimenai D, Watschinger B, Mariat C, Sever MS, Crespo M, Peruzzi L, Spasovski G, Sorensen SS, Heemann U, Pascual J, Viklicky O, Courtney AE, Hadaya K, Wagner L, Nistor I, Hadjianastassiou V, Durlik M, Helantera I, Oberbauer R, Oniscu G, Hilbrands L, Abramowicz D. Long-term risks after kidney donation: how do we inform potential donors? A survey from DESCARTES and EKITA transplantation working groups. Nephrol Dial Transplant. 2021 Aug 27;36(9):1742-1753. doi: 10.1093/ndt/gfab035. PMID 33585931
- [Background] Reichlin T, Twerenbold R, Reiter M, Steuer S, Bassetti S, Balmelli C, Winkler K, Kurz S, Stelzig C, Freese M, Drexler B, Haaf P, Zellweger C, Osswald S, Mueller C. Introduction of high-sensitivity troponin assays: impact on myocardial infarction incidence and prognosis. Am J Med. 2012 Dec;125(12):1205-1213.e1. doi: 10.1016/j.amjmed.2012.07.015. PMID 23164485
- [Background] Shah AS, Anand A, Sandoval Y, Lee KK, Smith SW, Adamson PD, Chapman AR, Langdon T, Sandeman D, Vaswani A, Strachan FE, Ferry A, Stirzaker AG, Reid A, Gray AJ, Collinson PO, McAllister DA, Apple FS, Newby DE, Mills NL; High-STEACS investigators. High-sensitivity cardiac troponin I at presentation in patients with suspected acute coronary syndrome: a cohort study. Lancet. 2015 Dec 19;386(10012):2481-8. doi: 10.1016/S0140-6736(15)00391-8. Epub 2015 Oct 8. PMID 26454362
- [Background] Chapman AR, Lee KK, McAllister DA, Cullen L, Greenslade JH, Parsonage W, Worster A, Kavsak PA, Blankenberg S, Neumann J, Sorensen NA, Westermann D, Buijs MM, Verdel GJE, Pickering JW, Than MP, Twerenbold R, Badertscher P, Sabti Z, Mueller C, Anand A, Adamson P, Strachan FE, Ferry A, Sandeman D, Gray A, Body R, Keevil B, Carlton E, Greaves K, Korley FK, Metkus TS, Sandoval Y, Apple FS, Newby DE, Shah ASV, Mills NL. Association of High-Sensitivity Cardiac Troponin I Concentration With Cardiac Outcomes in Patients With Suspected Acute Coronary Syndrome. JAMA. 2017 Nov 21;318(19):1913-1924. doi: 10.1001/jama.2017.17488. PMID 29127948
- [Background] Chapman AR, Anand A, Boeddinghaus J, Ferry AV, Sandeman D, Adamson PD, Andrews J, Tan S, Cheng SF, D'Souza M, Orme K, Strachan FE, Nestelberger T, Twerenbold R, Badertscher P, Reichlin T, Gray A, Shah ASV, Mueller C, Newby DE, Mills NL. Comparison of the Efficacy and Safety of Early Rule-Out Pathways for Acute Myocardial Infarction. Circulation. 2017 Apr 25;135(17):1586-1596. doi: 10.1161/CIRCULATIONAHA.116.025021. Epub 2016 Dec 29. PMID 28034899
- [Background] Kimenai DM, Janssen EBNJ, Eggers KM, Lindahl B, den Ruijter HM, Bekers O, Appelman Y, Meex SJR. Sex-Specific Versus Overall Clinical Decision Limits for Cardiac Troponin I and T for the Diagnosis of Acute Myocardial Infarction: A Systematic Review. Clin Chem. 2018 Jul;64(7):1034-1043. doi: 10.1373/clinchem.2018.286781. Epub 2018 May 29. PMID 29844245
- [Background] Apple FS, Ler R, Murakami MM. Determination of 19 cardiac troponin I and T assay 99th percentile values from a common presumably healthy population. Clin Chem. 2012 Nov;58(11):1574-81. doi: 10.1373/clinchem.2012.192716. Epub 2012 Sep 14. PMID 22983113
- [Background] Anand A, Shah ASV, Beshiri A, Jaffe AS, Mills NL. Global Adoption of High-Sensitivity Cardiac Troponins and the Universal Definition of Myocardial Infarction. Clin Chem. 2019 Mar;65(3):484-489. doi: 10.1373/clinchem.2018.298059. Epub 2019 Jan 9. PMID 30626631
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Wildi K, Gimenez MR, Twerenbold R, Reichlin T, Jaeger C, Heinzelmann A, Arnold C, Nelles B, Druey S, Haaf P, Hillinger P, Schaerli N, Kreutzinger P, Tanglay Y, Herrmann T, Moreno Weidmann Z, Krivoshei L, Freese M, Stelzig C, Puelacher C, Rentsch K, Osswald S, Mueller C. Misdiagnosis of Myocardial Infarction Related to Limitations of the Current Regulatory Approach to Define Clinical Decision Values for Cardiac Troponin. Circulation. 2015 Jun 9;131(23):2032-40. doi: 10.1161/CIRCULATIONAHA.114.014129. Epub 2015 May 6. PMID 25948541
- [Background] Kimenai DM, Gerritse BM, Lucas C, Rosseel PM, Bentala M, van Hattum P, van der Meer NJ, Scohy TV. Effectiveness of pericardial lavage with or without tranexamic acid in cardiac surgery patients receiving intravenous tranexamic acid: a randomized controlled trial. Eur J Cardiothorac Surg. 2016 Dec;50(6):1124-1131. doi: 10.1093/ejcts/ezw214. Epub 2016 Jun 21. PMID 27330150
- [Background] Mueller T, Egger M, Peer E, Jani E, Dieplinger B. Evaluation of sex-specific cut-off values of high-sensitivity cardiac troponin I and T assays in an emergency department setting - Results from the Linz Troponin (LITROP) study. Clin Chim Acta. 2018 Dec;487:66-74. doi: 10.1016/j.cca.2018.09.026. Epub 2018 Sep 15. PMID 30227114
- [Background] Ungerer JP, Marquart L, O'Rourke PK, Wilgen U, Pretorius CJ. Concordance, variance, and outliers in 4 contemporary cardiac troponin assays: implications for harmonization. Clin Chem. 2012 Jan;58(1):274-83. doi: 10.1373/clinchem.2011.175059. Epub 2011 Nov 28. PMID 22125306
- [Background] McDonald S, Furmuga J, Vigen R, et al. Assessment of agreement of two high sensitivity troponin assays during an institutional transition. Vessel Plus. 2021;5(38):1-8.
- [Background] Karady J, Mayrhofer T, Ferencik M, Nagurney JT, Udelson JE, Kammerlander AA, Fleg JL, Peacock WF, Januzzi JL Jr, Koenig W, Hoffmann U. Discordance of High-Sensitivity Troponin Assays in Patients With Suspected Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Mar 30;77(12):1487-1499. doi: 10.1016/j.jacc.2021.01.046. PMID 33766254
- [Background] Anand A, Lee KK, Chapman AR, Ferry AV, Adamson PD, Strachan FE, Berry C, Findlay I, Cruikshank A, Reid A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Harkess R, Keerie C, Weir CJ, Parker RA, Gray A, Shah ASV, Mills NL; HiSTORIC Investigatorsdagger. High-Sensitivity Cardiac Troponin on Presentation to Rule Out Myocardial Infarction: A Stepped-Wedge Cluster Randomized Controlled Trial. Circulation. 2021 Jun 8;143(23):2214-2224. doi: 10.1161/CIRCULATIONAHA.120.052380. Epub 2021 Mar 23. PMID 33752439
- [Derived] Boeddinghaus J, Li Z, Bularga A, Taggart C, Wereski R, Chapman AR, Lee KK, Tuck C, Gunn R, Jenks S, McCance K, Pattenden R, Malo J, Thurston AJF, Tew YY, McDermott M, Gray A, Cruden NLM, Anand A, Kimenai DM, Mills NL; TWITCH-ED Investigators. Clinical Decisions and Outcomes After Switching High-Sensitivity Cardiac Troponin Assays in Suspected ACS: An Interrupted Time-Series Study. JAMA Cardiol. 2025 Dec 17:e254661. doi: 10.1001/jamacardio.2025.4661. Online ahead of print. PMID 41405901